CLINICAL TRIAL: NCT07130786
Title: A Phase II Randomized Open-Label Trial of Levetiracetam for Prevention of Seizures in Patients With Brain Metastases in Primary Motor Cortex
Brief Title: Prophylactic Anti-Seizure Medication vs No Anti-Seizure Medication for Patients With Primary Motor Cortex Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ayal A. Aizer, MD (Other)
Responsible Party: Sponsor-Investigator, Ayal A. Aizer, MD, Director, Central Nervous System Radiation Oncology; Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-189
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Seizures; Primary Motor Cortex; Brain Metastases From Non-small Cell Lung Cancer (NSCLC); Brain Metastases, Adult; Brain Metastases From Extra-cranial Solid Tumors
Keywords: brain metastases; seizure; levetiracetam; seizure-naive; keppra; motor; primary motor cortex; motor strip; prophylaxis; Anti-Seizure Medication; ASM; SRS; SRT; necrosis; local recurrence; quality of life; focal aware; focal impaired awareness; focal to bilateral tonic clonic; generalized; focal preserved consciousness; focal impaired consciousness; FPC; FIC; FTBC; tonic; clonic
MeSH Terms: conditions — Seizures; Brain Neoplasms; Necrosis | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prophylactic Levetiracetam (Experimental): Levetiracetam Anti-Seizure Medication
  Interventions: Drug: Levetiracetam (Keppra)
- No Prophylactic Levetiracetam (No Intervention): No Anti-Seizure Medication

INTERVENTIONS:
Drug: Levetiracetam (Keppra) — Patients will be randomized to receive levetiracetam/ASM or to receive no ASM therapy
  Arms: Prophylactic Levetiracetam

SUMMARY:
This is a randomized trial for patients with brain metastases in the primary motor cortex who have not had seizures to receive either the prophylactic anti-seizure medication levetiracetam (also known by its trade name Keppra) or proceed with standard of care management, which does not currently include prophylactic levetiracetam. Patients who enroll to this trial will be randomized to receive prophylactic levetiracetam or not receive prophylactic levetiracetam.

DETAILED DESCRIPTION:
Brain metastases (BrM) impact 10%-40% of patients with solid malignancies and are associated with significant clinical sequelae, including development of seizures. The development of seizures has the potential for significant detriment on patient quality of life. The goal of this study is to evaluate the role of levetiracetam as primary prophylaxis in seizure-naïve patients with metastases in primary motor cortex, an area at high risk of seizures. Patients will be randomized to receive levetiracetam/ASM or to receive no ASM therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a biopsy proven solid malignancy with at least one intracranial lesion radiographically consistent with or pathologically proven to be a brain metastasis located in the primary motor cortex measuring 0.5 cm or larger in maximal unidimensional size
2. Age of at least 18 years
3. Karnofsky performance status of at least 60
4. Estimated survival of at least 3-6 months in the opinion of the enrolling clinician and/or study PI
5. Ability to understand and the willingness to sign a written informed consent document by either ink on paper or a DF/HCC approved eConsent medium

Exclusion Criteria:

1. Participants with prior seizures as this is a study for seizure naïve patients
2. Participants with an allergy to levetiracetam as levetiracetam is the prophylactic anti-seizure medication under study
3. Participants concurrently taking (i.e. at enrollment) an ASM for non-seizure indications at clinically relevant doses (gabapentin 1800 mg/day or higher, pregabalin 300 mg/ day or higher, lamotrigine 150 mg/ day or higher, valproic acid 1000 mg/ day or higher, topiramate 200 mg/ day or higher, carbamazepine 200 mg/ day or higher, oxcarbazepine 300 mg/ day or higher, primidone 100 mg/day or higher) because use of these medications could bias the study toward the null
4. Participants who cannot tolerate a magnetic resonance imaging (MRI) study of the brain, which is required to determine the presence of and follow the course of brain metastases under study
5. Participants who cannot receive gadolinium as MRI of the brain with contrast is required
6. Participants with end stage renal disease due to risk of nephrogenic systemic fibrosis in this patient population after exposure to gadolinium-based contrast agents
7. Participants with widespread, definitive leptomeningeal disease given that leptomeningeal disease and brain metastases are different entities
8. Pregnant women are excluded from this study because levetiracetam crosses the placenta. In addition, the potential deleterious effects of gadolinium on the developing fetus are not completely known
9. Women who are breastfeeding are excluded from this study because levetiracetam enters breast milk. In addition, the potential deleterious effects of gadolinium in breast milk remain unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Seizure Rate | Duration of time on study (estimated 1 year)
  To determine whether seizure rate is lower in seizure-naïve patients with brain metastases in primary motor cortex with levetiracetam prophylaxis versus usual care of no ASM therapy.

SECONDARY OUTCOMES:
Overall survival | Duration of time on study (estimated 1 year)
  Clinical parameter
Death due to neurologic disease progression | Duration of time on study (estimated 1 year)
  Clinical parameter to be assessed via review of study visits and medical records indicating cause of death (neurologic versus non-neurologic)
Progression free survival | Duration of time on study (estimated 1 year)
  Clinical assessment time to first progression after baseline
Performance status | Duration of time on study (estimated 1 year)
  Karnofsky performance status (KPS). Assessed longitudinally. Higher scores on 0-100 scale represent better functional status and less dependence on others.
Time to detection of new brain metastases | Duration of time on study (estimated 1 year)
  Radiographic assessment showing first appearance of new brain metastases after baseline
Time to development of radiation necrosis | Duration of time on study (estimated 1 year)
  Radiographic assessment of first appearance of radiation necrosis after baseline
Time to development of leptomeningeal disease | Duration of time on study (estimated 1 year)
  Radiographic assessment of first appearance of leptomeningeal disease after baseline
Time to local recurrence | Duration of time on study (estimated 1 year)
  Radiographic assessment of first local recurrence after baseline in brain metastases treated with radiation
Time to craniotomy | Duration of time on study (estimated 1 year)
  Clinical assessment of first use of neurosurgical resection as salvage therapy after baseline
Time to radiotherapeutic treatments after initial management | Duration of time on study (estimated 1 year)
  Clinical assessment of first use of salvage brain-directed radiation after baseline
Quality of life/symptom burden and interference | Duration of time on study (estimated 1 year)
  Questionnaire - MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) - Items assessed on a 0-10 scale with 10 being the highest severity. Cumulative scores with higher values reflect greater interference/severity of symptoms.
  Assessed longitudinally.
  Questionnaire - Quality of Life in Epilepsy Inventory - 31(QOLIE-31)
  - Final score from 0-100 with higher scores reflecting greater quality of life. Higher T scores similarly reflect greater quality of life.
  Assessed longitudinally.
Seizure type | Duration of time on study (estimated 1 year)
  Clinical determination of type of seizure (if present) after baseline. Type of seizure: focal preserved consciousness, focal impaired consciousness, focal to bilateral-tonic-clonic, each adjudicated with or without observable manifestations and with semiology incorporated including elementary motor phenomena
Time to seizure | Duration of time on study (estimated 1 year)
  Time to clinical determination of presence of primary seizure after baseline
Seizure rate in the week following brain-directed local therapy such as brain-directed surgery or radiation | Duration of time on study (estimated 1 year)
  Clinical determination of presence and number of seizure(s) in the week following brain-directed surgery or radiation after baseline
Time to secondary seizures | Duration of time on study (estimated 1 year)
  Clinical determination of presence of secondary seizures after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ayal A Aizer, MD, MHS, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided